CLINICAL TRIAL: NCT07325422
Title: Weizmannia Coagulans BC99 Relieves Exercise-induced Fatigue: a Randomized Controlled Trial
Brief Title: Weizmannia Coagulans BC99 Relieves Exercise-induced Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20251226
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: College Student

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): 3g dose of milk protein concentrate/pack, 8 packs per day
  Interventions: Dietary Supplement: Placebo
- BC99 group (Experimental): 3g dose of milk protein concentrate with 6×109 Colony Forming Unit (CFU) W. coagulans BC99/pack, 8 packs per day
  Interventions: Dietary Supplement: BC99

INTERVENTIONS:
Dietary Supplement: Placebo — The experimental phase of this study lasts 12 weeks and each subject will have 3 visits (Week 0, Week 6, Week 12)
  Arms: Placebo group
Dietary Supplement: BC99 — The experimental phase of this study lasts 12 weeks and each subject will have 3 visits (Week 0, Week 6, Week 12)
  Arms: BC99 group

SUMMARY:
To evaluate the clinical effects of Weizmannia coagulans BC99 supplementation compared with placebo on plasma amino acid profiles in male university students following a 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19-35 years, with no restriction on sex;
2. Physically active individuals with regular daily exercise training intensity and duration;
3. No history of allergy to protein products;
4. Body weight ≥50 kg for male subjects and ≥45 kg for female subjects; body mass index (BMI), calculated as weight (kg) divided by height squared (m²), within the range of 19.0-24.0 kg/m²;
5. No history of cardiovascular or cerebrovascular diseases, hypertension, diabetes, hepatic or renal dysfunction, or other underlying diseases or metabolic disorders;
6. Willingness to comply with the study protocol and study restrictions, and voluntary provision of written informed consent to participate in the study.

Exclusion Criteria:

1. History of allergic constitution or immunodeficiency;
2. Blood donation or significant blood loss (≥200 mL) within 3 months prior to administration of the investigational product;
3. Presence of severe diseases of major organs, including the cardiovascular system, lungs, liver, or kidneys, as well as diabetes mellitus, severe thyroid disorders, metabolic diseases, malignant tumors, or severe immune system diseases;
4. Use of medications affecting the intestinal microbiota (including antibiotics, microecological preparations, intestinal mucosal protectants, traditional Chinese medicines, etc.) for more than one consecutive week within 1 month prior to screening;
5. Any other condition that, in the investigator's judgment, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Changes of amino acids | 12 weeks
  Plasma amino acid changes were determined by targeted UHPLC-MS/MS analysis using isotope-labeled internal standards and quality control samples to ensure analytical accuracy and reproducibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Wu Ying, Luoyang, Henan, China